CLINICAL TRIAL: NCT04679844
Title: A Prospective, Randomized, Multi-Center Study to Assess the Safety and Performance of MagnetOs Easypack Putty Standalone Compared to Demineralized Bone Matrix or Fibers (DBX or Grafton) Mixed With Local Autograft in Patients Undergoing One to Two-Level Instrumented Posterolateral Lumbar/Thoracolumbar Fusion (PLF)
Brief Title: Post Marketing Study of MagnetOs Easypack Putty Standalone Compared to Demineralized Bone Matrix or Fibers Mixed With Autograft in Patients Undergoing Posterolateral Lumbar Fusion
Acronym: PROOF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuros Biosurgery AG (Industry)
Collaborators: Simplified Clinical Data Systems, LLC (Industry); Kuros BioSciences B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAG-920-023
Record Dates: First submitted 2020-12-18; First posted 2020-12-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Degenerative Disc Disease; Spine Fusion; Back Pain
Keywords: Degenerative Disc Disease; Spine Fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration; Back Pain

STUDY DESIGN:
Intervention Model Description: Intra-patient control. Each patient serves as their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MagnetOs Easypack Putty (Experimental): Interventions
  * Procedure: Instrumented posterolateral spine fusion
  * Device; MagnetOs Easypack Putty
  Interventions: Device: MagnetOs Easypack Putty
- Demineralized Bone Matrix or Fibers (DBX or Grafton) mixed with local autograft bone (Active Comparator): Interventions
  * Procedure: Instrumented posterolateral spine fusion
  * Device: Demineralized Bone Matrix or Fibers mixed with local autograft bone
  Interventions: Device: Demineralized Bone Matrix or Fibers mixed with local autograft bone

INTERVENTIONS:
Device: MagnetOs Easypack Putty — MagnetOs Easypack Putty used standalone in instrumented posterolateral fusion, 5cc-15c per spine level at the randomized assigned side.
  Arms: MagnetOs Easypack Putty
Device: Demineralized Bone Matrix or Fibers mixed with local autograft bone — Demineralized Bone Matrix or Fibers (DBX or Grafton) mixed in a 1:1 vol% with local autologous bone graft used in instrumented posterolateral fusion, 5cc-15cc per level mixed with bone marrow aspirate/blood per spine level at the contralateral side.
  Arms: Demineralized Bone Matrix or Fibers (DBX or Grafton) mixed with local autograft bone

SUMMARY:
This is a phase IV post-marketing study for MagnetOs Easypack Putty. MagnetOs Easypack Putty is a synthetic bone graft extender product that is routinely used by surgeons as a treatment for patients with degenerative disc disease or spinal trauma undergoing spinal fusion surgery.

In this study, MagnetOs Easypack Putty will be used according to the latest U.S. Instructions For Use, standalone in the posterolateral spine.

DETAILED DESCRIPTION:
In this study, following a screening period of a maximum of 30 days, 60 patients will undergo up to two-level instrumented posterolateral fusion (PLF) procedure. Prior to surgery, each patient will be randomized to receive MagnetOs Easypack Putty standalone on the assigned side of the spine and Demineralized Bone Matrix or Fibers mixed with local autograft bone on the other at the diseased levels. They will be followed up at discharge, Week 2, Month 3, Month 6, and Month 12. An interim analysis will be performed once 30 patients have completed their Month 6 visit and have measurements for the endpoints available to measure effectiveness. The primary endpoint will be analyzed at Month 12.

In this study, MagnetOs Easypack Putty will be applied according to the latest Instructions for Use approved in the United States. Specifically, MagnetOs Easypack Putty will be used standalone in patients up to two-level degenerative disc disease with segmental mechanical spinal instability requiring treatment with an instrumented posterolateral spine fusion procedure. The fusion procedure (PLF) will be left to the surgeon's discretion.

Radiographs will be obtained at Screening, Discharge, Month 3, Month 6 and Month 12. CT scans will only be obtained at Month 6 and Month 12.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to read/be read, understand, and provide written informed consent and has signed the Institutional Review Board (IRB) approved informed consent.
* Male or female patient ≥ 18 years old.
* Patients with segmental mechanical spinal instability requiring arthrodesis surgery.

Instability can be either caused by degenerative disc disease or by traumatic injury to the spinal column. Patient requiring a maximum of two-level instrumented posterolateral lumbar/thoraco-lumbar fusion (T11 - S1) will be enrolled. Mechanical instability is defined by the presence of one or more of the following:

1. instability (angulation ≥ 5 degrees or translation ≥ 3 mm on flexion/extension radiographs),
2. decreased disc height by > 2 mm, but dependent upon the spinal level
3. Grade II or more listhesis
4. TLICS equal or greater than 5
5. Unstable burst fracture

   * Failed conservative treatment (physical therapy, bed rest, medications, spinal injections, manipulations, or transcutaneous electrical nerve stimulation) for a minimum period of 3 months prior to study enrollment (if the patient undergoes elective surgery). Patients who have spinal instability (as defined above in inclusion criteria number three), caused by acute trauma requiring urgent surgical treatment are excluded from this criterion.

Exclusion Criteria:

* Requires > two-level fusion or expected to need secondary intervention within one year following surgery.
* Had prior PLF fusion or attempted PLF fusion at the involved levels.
* Had previous decompression at the involved levels.
* Women who are or intend to become pregnant within the next 12 months.
* To treat conditions in which general bone grafting is not advisable.
* In conditions where the surgical site may be subjected to excessive impact or stresses, including those beyond the load strength of fixation hardware (e.g. defect site stabilization is not possible).
* In case of significant vascular impairment proximal to the graft site.
* In case of severe metabolic or systemic bone disorders (e.g., osteogenesis imperfecta, history of or active Pott's disease, stage >4 renal disease or Paget's Disease) that affect bone or wound healing.
* In case of acute and chronic infections in the operated area (soft tissue infections; inflammation, bacterial bone diseases; osteomyelitis).
* When intraoperative soft tissue coverage is not planned or possible.
* Receiving treatment with medication interfering with calcium metabolism.
* Has degenerative disc disease (DDD) related to a benign or malignant tumor.
* Has history or presence of active malignancy.
* Has known substance abuse, psychiatric disorder, or a condition which, in the opinion of the investigator, may influence the healing or ability to comply with protocol requirements.
* Is involved in active litigation relating to his/her spinal condition.
* Has participated in an investigational study within 30 days prior to surgery for study devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2027-06-02 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic Fusion by CT Scan | Month 12
  The rate of posterolateral lumbar/thoracolumbar fusion assessed by CT-scan at Month 12. Radiographic as determined by evidence of bridging trabeculae or continuous bony connection between the superior and inferior transverse processes.

SECONDARY OUTCOMES:
Radiographic Fusion by Plain Radiographs | Month 6, Month 12
  The rate of posterolateral lumbar/thoracolumbar fusion assessed by plain radiographs.
Radiographic Fusion by CT Scan | Month 6
  The rate of posterolateral lumbar/thoracolumbar fusion assessed by CT-scan at Month 6. Radiographic as determined by evidence of bridging trabeculae or continuous bony connection between the superior and inferior transverse processes.
Functional Outcome by Oswestry Disability Index Questionnaire | Screening, Week 2, Month 3, 6, and 12
  Functional outcome by the Oswestry Disability Index questionnaire. Patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain. The lower the percentage the higher the patient's functionality. 0-20% minimal disability, 80-100% significant disability or bedridden.
Back and Leg Pain by Visual Analog Pain Scale Questionnaire | Screening, Week 2, Month 3, 6, and 12
  Change in back and leg pain using Visual Analog Pain Scale (0-100). Patient-completed questionnaire scoring pain by using 100 mm line. Zero being no pain, 100 is worst pain imaginable.
Neurologic Status by Physical Exam | Screening, Week 2, Month 3, 6, and 12
  Change in neurologic status by examination to document stable, improved, or deficits in condition. Stable or improved findings for lower extremities, specifically reflexes, muscle strength, sensory, and straight leg raise.
Success Rate | Week 2, Month 3, 6, and 12
  Number of patients with secondary surgical interventions (SSI's) such as revisions, re-operations, removals, supplemental fixations, or any other procedure that adjusts or removes part of the original implant configuration with or without replacement of the components within 12 months of surgery.

OTHER OUTCOMES:
Safety Endpoint - number of patients with Adverse Events | 12 Months
  The number of patients with Adverse Events from Screening up to Month 12 after surgery.
Safety Endpoint - number of patients with Serious Adverse Events | 12 Months
  The number of patients with Serious Adverse Events from Screening up to Month 12 after surgery
Safety Endpoint - number of patients with Adverse Device Effects | 12 Months
  The number of patients with Adverse Device Effects from Screening up to Month 12 after surgery.
Safety Endpoint - number of patients with Device Related Complications | 12 Months
  The number of patients with any complications considered to device related with 12 months after surgery.
Health Economic - Duration of Surgery | 12 Months
  Duration of surgery in minutes.
Health Economic - Duration of Hospitalization | 12 Months
  Duration of hospital stay in days.
Health Economic - Return to Work | 12 Months
  Time to return to work in days.

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Silva, MD, Study Director — Kuros BioSciences B.V.
Locations (4):
- United States (4):
  - The Washington University, St Louis, Missouri
  - Rothman Orthopaedic Institute, Philadelphia, Pennsylvania
  - Tennessee Orthopaedic Alliance, Nashville, Tennessee
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No